CLINICAL TRIAL: NCT04104256
Title: Pragmatic Trial of an Electronic Health Record/Behavioral Economics Intervention to Reduce Pre-Operative Testing for Cataract Surgery
Brief Title: Using Behavioral Economics to Reduce Low-Value Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: RAND (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01AG059815-01 (NIH); 5R01AG059815 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pre-Operative Testing for Cataract Surgery
Keywords: Low Value Care; Cataract Surgery; Behavioral Economics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alert 1 (Experimental): Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #1 group.
  Interventions: Behavioral: Nudge #1: Alert highlighting the safety/potential harms to patients of undergoing pre-op tests
- Alert 2 (Experimental): Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #2 group.
  Interventions: Behavioral: Nudge #2: Alert highlighting the financial harms to the patient experiencing pre-op tests
- Alert 3 (Experimental): Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #3 group.
  Interventions: Behavioral: Nudge #3: Alert highlighting potential psychological harms to the patient of experiencing pre-op tests
- Control (Experimental): Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Control group. Encounter continues as usual.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Nudge #1: Alert highlighting the safety/potential harms to patients of undergoing pre-op tests — Nudge 1:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-op tests do NOT increase patient safety and go AGAINST local and national guidelines Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
  Arms: Alert 1
Behavioral: Nudge #2: Alert highlighting the financial harms to the patient experiencing pre-op tests — Nudge #2:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can increase the patient's out-of-pocket costs without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Nudge includes "hard stop" before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
  Arms: Alert 2
Behavioral: Nudge #3: Alert highlighting potential psychological harms to the patient of experiencing pre-op tests — Nudge 3:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can cause aggravation and psychological stress for the patient without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
  Arms: Alert 3
Other: Usual Care — Patients will receive usual care from their physicians.
  Other Names: Control
  Arms: Control

SUMMARY:
There is strong consensus - based on robust randomized trial data - that routine pre-operative (pre-op) testing for cataract surgery is inappropriate. Despite these widely endorsed evidence-based recommendations, most seniors undergoing cataract surgery still receive unnecessary blood testing, EKGs, and chest X-rays (CXRs); another substantial percentage even undergo nonindicated cardiac stress tests. We will integrate three new best practice alert (BPA) nudges into the University of California, Los Angeles (UCLA) Health electronic health record (EHR). The nudges are informed by behavioral economic theory and are designed to alter the choice architecture for physicians to decrease the rate of pre-op test ordering while still preserving clinician autonomy. We will conduct a pragmatic trial to evaluate whether these BPA nudges reduce low-value pre-op testing for cataract surgery.

DETAILED DESCRIPTION:
There is strong consensus - based on robust randomized trial data - that routine pre-operative (pre-op) testing for cataract surgery is inappropriate (Keay et al, 2009; Keay et al, 2012; Schein et al, 2000; Chen et al, 2015). Because pre-op testing provides no benefit to patients, the American Academy of Ophthalmology named reducing routine pre-op testing for cataract surgery the #1 issue that patients and physicians should question as part of the Choosing Wisely™ campaign (Schein et al, 2012). Despite these widely endorsed evidence-based recommendations, most seniors undergoing cataract surgery still receive unnecessary blood testing, EKGs, and chest X-rays (CXRs); another substantial percentage even undergo non-indicated cardiac stress tests (Rumball-Smith et al, 2017).

With cataract surgery being the most common medical procedure among Medicare beneficiaries (predicted 4.4 million per year by the year 2030) (Schein et al, 2012), widespread reduction of routine pre-op testing for cataract surgery would reduce costs, reduce exposure to unnecessary and potentially harmful tests, and allow millions of seniors to spend more time enjoying life rather than wasting their time receiving inappropriate health care.

The investigators hypothesize that an interdisciplinary electronic health record (EHR)-based intervention that applies behavioral economics approaches (i.e., "nudges") will dramatically reduce pre-op testing for cataract surgery in a real-world clinical setting. The investigators propose to test this hypothesis by conducting a pragmatic randomized trial, implementing this intervention at UCLA Health (Ronald Reagan UCLA Medical Center), where ~3200 cataract surgeries are performed per year. The specific aims are to:

1. Integrate three new BPA nudges into the UCLA Health EHR. The investigators will conduct a four-arm randomized pragmatic trial to compare the effectiveness of the nudges vs. usual care. Three distinct nudges were tailored to highlight the safety aspects of pre-op tests, the financial harms to the patient of experiencing pre-op tests, and the potential psychological harms to the patient of experiencing preop tests. The pragmatic trial will include three types of behavioral nudges to promote the desired reduction in low value care:

   Nudge 1:
   * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
   * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
   * Routine pre-op tests are inappropriate.
   * Routine pre-op tests do NOT increase patient safety and go AGAINST local and national guidelines
   * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"

   Nudge 2:
   * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
   * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
   * Routine pre-op tests are inappropriate.
   * Routine pre-operative tests can increase the patient's out-of-pocket costs without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
   * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"

   Nudge 3:
   * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
   * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
   * Routine pre-op tests are inappropriate.
   * Routine pre-operative tests can cause aggravation and psychological stress for the patient without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
   * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
2. Randomize providers who conducted a pre-op visit in 2019 and those who are expected to conduct such a visit during the 12-month study period to one of 4 study arms (usual pre-op care, Nudge #1, Nudge #2, or Nudge #3) and measure and compare the efficacy of each intervention. The investigators will measure and compare rates of testing before and after initiation of the randomization. Outcomes will be measured 12-months after the intervention start date.

For the primary outcome, we will assess the change in the percentage of cataract patients who undergo one or more pre-op tests after 12 months, where the baseline comparison will be 2019. While we intended to the 12-month pre-period as the baseline, the COVID-19 pandemic had a substantial impact on cataract surgeries. We will compare the percentage of patients receiving pre-op testing in the pooled nudge arms to the usual care arm (primary outcome) and measure the efficacy of each individual nudge arm to determine whether certain behavioral economic framing techniques are more effective than others at reducing pre-op testing (secondary outcomes). Other secondary outcomes will include the change in the percentage of patients who received pre-op labs, pre-op EKGs, and pre-op CXRs. We will also evaluate the total number of pre-op tests patients received, same-day surgery cancellations, cost savings to the health system, and cost savings to the patient. To elicit the views and experiences of physicians, we will survey physicians randomized to all intervention arms to evaluate their experience with the EHR alerts.

Reducing patient exposure to unnecessary care is central to improving patient outcomes and value. This project is fully aligned with UCLA Health leadership's current priority of supporting cross-departmental system change to improve quality of care, outcomes, and value for UCLA patients. Because of the close partnership between our UCLA Informatics co-Investigators and the EHR vendor (Epic), the low-cost intervention that we propose to implement and test will be easily disseminatable to all Epic-based health systems, and will have the potential to dramatically reduce inappropriate pre-op testing across the nation.

EHRs are in their infancy, and the scientific community is only beginning to learn how to use them as tools to promote desired care processes (Meeker et al, 2016). This proposed pragmatic trial would break new ground in our understanding of how behavioral economics approaches can be used to tamp down on care that does not promote better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient at UCLA undergoing cataract surgery, and receives pre-operative evaluation at UCLA Health

Exclusion Criteria:

* Cataract surgery patients who get their pre-operative evaluation from non-UCLA physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Sarkisian, MD, MSPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keay L, Lindsley K, Tielsch J, Katz J, Schein O. Routine preoperative medical testing for cataract surgery. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007293. doi: 10.1002/14651858.CD007293.pub2. PMID 19370681
- [Background] Keay L, Lindsley K, Tielsch J, Katz J, Schein O. Routine preoperative medical testing for cataract surgery. Cochrane Database Syst Rev. 2012 Mar 14;3(3):CD007293. doi: 10.1002/14651858.CD007293.pub3. PMID 22419323
- [Background] Schein OD, Katz J, Bass EB, Tielsch JM, Lubomski LH, Feldman MA, Petty BG, Steinberg EP. The value of routine preoperative medical testing before cataract surgery. Study of Medical Testing for Cataract Surgery. N Engl J Med. 2000 Jan 20;342(3):168-75. doi: 10.1056/NEJM200001203420304. PMID 10639542
- [Background] Chen CL, Lin GA, Bardach NS, Clay TH, Boscardin WJ, Gelb AW, Maze M, Gropper MA, Dudley RA. Preoperative medical testing in Medicare patients undergoing cataract surgery. N Engl J Med. 2015 Apr 16;372(16):1530-8. doi: 10.1056/NEJMsa1410846. PMID 25875258
- [Background] Schein OD, Cassard SD, Tielsch JM, Gower EW. Cataract surgery among Medicare beneficiaries. Ophthalmic Epidemiol. 2012 Oct;19(5):257-64. doi: 10.3109/09286586.2012.698692. PMID 22978526
- [Background] Rumball-Smith J, Shekelle PG, Bates DW. Using the Electronic Health Record to Understand and Minimize Overuse. JAMA. 2017 Jan 17;317(3):257-258. doi: 10.1001/jama.2016.18609. No abstract available. PMID 28114561
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Derived] Ahmadi A, Sorensen A, Villaflores CWA, Mafi JN, Vangala SS, Hofer IS, Bartlett JD, Cheng EM, Duval VF, Damberg C, Elashoff D, Goldstein NJ, Ladapo JA, Moore JM, Pessegueiro AM, Shu SB, Skootsky SA, Turner A, Sarkisian CA. Protocol for pragmatic randomised trial: integrating electronic health record-based behavioural economic 'nudges' into the electronic health record to reduce preoperative testing for patients undergoing cataract surgery. BMJ Open. 2021 Nov 3;11(11):e049568. doi: 10.1136/bmjopen-2021-049568. PMID 34732478
- See also: Choosing Wisely®. American Academy of Ophthalmology: Five Things Physicians and Patients Should Question. 2013 — http://www.choosingwisely.org/societies/american-academy-of-ophthalmology/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled into the study when they have a pre-operative encounter for cataract surgery AND the physician starts to order a pre-op lab. Eligible providers were assigned an arm of the study based on their 2019 pre-operative visits. Patients were enrolled into each arm based on the providers arm assignment. Healthcare Providers were not enrolled in the study
Groups:
- Alert 1: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #1 group.
  Nudge #1: Alert highlighting the safety/potential harms to patients of undergoing pre-op tests: Nudge 1:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-op tests do NOT increase patient safety and go AGAINST local and national guidelines Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
- Alert 2: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #2 group.
  Nudge #2: Alert highlighting the financial harms to the patient experiencing pre-op tests: Nudge #2:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can increase the patient's out-of-pocket costs without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Nudge includes "hard stop" before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
- Alert 3: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #3 group.
  Nudge #3: Alert highlighting potential psychological harms to the patient of experiencing pre-op tests: Nudge 3:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can cause aggravation and psychological stress for the patient without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
Period: Overall Study
Arm/Group | Alert 1 | Alert 2 | Alert 3 | Control
Started | 269 | 267 | 272 | 237
Completed | 269 | 267 | 272 | 237
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Providers were not assessed for baseline
Groups:
- Alert 2: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #2 group
  Nudge #2: Alert highlighting the financial harms to the patient experiencing pre-op tests: Nudge #2:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can increase the patient's out-of-pocket costs without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Nudge includes "hard stop" before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
- Alert 3: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #3 group
  Nudge #3: Alert highlighting potential psychological harms to the patient of experiencing pre-op tests: Nudge 3:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-operative tests can cause aggravation and psychological stress for the patient without improving the safety or medical outcomes of cataract surgery and go AGAINST local and national guidelines
  * Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
- Control: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Control group.
  Usual Care: Patients will receive usual care from their physicians.
- Total: Total of all reporting groups
Arm/Group | Alert 1 | Alert 2 | Alert 3 | Control | Total
Number analyzed (Participants) | 269 | 267 | 272 | 237 | 1045
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.07 (9.58) | 72.00 (10.98) | 72.98 (9.61) | 72.27 (10.24) | 72.08 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 140 | 161 | 126 | 595
  Male | 101 | 127 | 111 | 111 | 450
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 34 | 38 | 26 | 126
  Not Hispanic or Latino | 214 | 203 | 204 | 178 | 799
  Unknown or Not Reported | 27 | 30 | 30 | 33 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  EthnoRacial Category: Black or African American | 20 | 11 | 18 | 18 | 67
  EthnoRacial Category: White | 142 | 132 | 148 | 131 | 553
  EthnoRacial Category: Unknown or Not Reported | 36 | 40 | 29 | 30 | 135
  EthnoRacial Category: Asian | 33 | 45 | 31 | 24 | 133
  EthnoRacial Category: Hispanic or Latino | 26 | 32 | 37 | 26 | 121
  EthnoRacial Category: Middle Eastern or North African | 7 | 4 | 5 | 5 | 21
  EthnoRacial Category: Multiple Ethnoracial Categories | 5 | 3 | 3 | 2 | 13
  EthnoRacial Category: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pre-Operative Testing Change
Description: Change in percentage of patients undergoing pre-operative testing (labs, EKG, CXR)
Time Frame: Pre-intervention (Baseline), Post-Intervention (12 months)
Population: The participants in this study are UCLA Health physicians who complete a pre-op visit for at least one patient undergoing cataract surgery at UCLA in the 12 months prior and 12 months after the study start date and all patients who are seen during such visits.
Measure: Mean (Standard Deviation); unit: Percentage of patients with orders
Groups:
- Control: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Control group
  Usual Care: Patients will receive usual care from their physicians.
Arm/Group | Alert 1 | Alert 2 | Alert 3 | Control
Number analyzed (Participants) | 75 | 66 | 69 | 76
Percentage of patients with orders
  Pre | 87.4 (33.2) | 85.0 (35.8) | 86.1 (34.6) | 85.4 (35.4)
  Post | 84.6 (36.2) | 80.3 (39.9) | 79.8 (40.3) | 83.5 (37.2)

2. Secondary Outcome: Pre-Operative Testing Change
Description: Efficacy of each individual nudge arm compared with usual care to determine whether certain behavioral economic framing techniques are more effective than others at reducing pre-op testing.
Time Frame: Pre-intervention (Baseline), Post-Intervention (12 months)
Reporting Status: Not Posted

3. Secondary Outcome: Pre-Operative Testing Change for Specific Categories of Tests
Description: Change in the percentage of patients who received pre-op labs, pre-op EKGs, and pre-op chest x-rays (CXRs).
Time Frame: Pre-intervention (Baseline), Post-Intervention (12 months)
Reporting Status: Not Posted

4. Secondary Outcome: Physician Experience Survey Results
Description: Perceived change in workflow, autonomy, satisfaction (Modified Survey)
Time Frame: Post-Intervention (12 months)
Reporting Status: Not Posted

5. Secondary Outcome: System-level Change - Surgery Cancellations
Description: Analysis of day of surgery cancellations for enrolled participants
Time Frame: Baseline, 12 months
Reporting Status: Not Posted

6. Secondary Outcome: System-level Change - Cost Savings
Description: Analysis of costs saved for enrolled participants
Time Frame: Pre-intervention (Baseline), Post-Intervention (12 months)
Reporting Status: Not Posted

7. Secondary Outcome: System-level Change - Return on Investment
Description: Analysis of cost savings to the health system assuming a reduction of tests being ordered
Time Frame: Pre-intervention (Baseline), Post-Intervention (12 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Post-Intervention (3 Months) Patients were monitored for the completion of their cataract surgery following their pre-op visit. Adverse events were then monitored/assessed for 12 weeks following the completion of their cataract surgery.
Description: An adverse event is defined as an Emergency Department visit that did not require hospitalization.
  Serious adverse events include hospitalization or death.
  Providers were not assessed for adverse events
Groups:
- Alert 1: Patients with a pre-op encounter in which the physician attempts to place an order for a pre-op test. Physician has been assigned to the Nudge #1 group
  Nudge #1: Alert highlighting the safety/potential harms to patients of undergoing pre-op tests: Nudge 1:
  * UCLA Ophthalmologists and Anesthesiologists ADVISE AGAINST routine pre-op testing.
  * UCLA Pre-op Eval and Planning Center (PEPC) will order any needed labs on the day of surgery.
  * Routine pre-op tests are inappropriate.
  * Routine pre-op tests do NOT increase patient safety and go AGAINST local and national guidelines Hard stop before allowing the ordering of a pre-op test where physicians must provide accountable justification: "EXPLAIN WHY GOING AGAINST GUIDELINES"
Arm/Group | Alert 1 | Alert 2 | Alert 3 | Control
All-Cause Mortality (participants affected / at risk) | 1/269 | 3/267 | 0/272 | 2/237
Serious Adverse Events (participants affected / at risk) | 11/269 | 4/267 | 4/272 | 12/237
Other Adverse Events (participants affected / at risk) | 9/269 | 7/267 | 12/272 | 12/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alert 1 (N=269) | Alert 2 (N=267) | Alert 3 (N=272) | Control (N=237)
Inpatient Admission (General disorders) | 11 | 4 | 4 | 12 — All inpatient admissions of enrolled participants were chart reviewed when admitted up to 12 weeks following cataract surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alert 1 (N=269) | Alert 2 (N=267) | Alert 3 (N=272) | Control (N=237)
Emergency Department visits that did not require admissions (General disorders) | 9 | 7 | 12 | 12 — All emergency department visits of enrolled participants were chart reviewed when emergency department visit occurred up to 12 weeks following cataract surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04104256/Prot_SAP_000.pdf